CLINICAL TRIAL: NCT00741351
Title: Anesthesiological Strategies in Elective Craniotomy: Randomized, Equivalence, Open Trial
Brief Title: Anesthesiological Strategies in Elective Craniotomy
Acronym: Neuromorfeo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Dott. Giuseppe Citerio, MD, Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT number 2007-005279-32; AIFA FARM6FKJKK
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Anesthesia; Craniotomy; Neurosurgery
Keywords: Anesthesia; Craniotomy; Neurosurgery
MeSH Terms: interventions — Sevoflurane; Fentanyl; Remifentanil; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IF (Experimental): Sevoflurane (Inhalation)+Fentanyl
  Interventions: Drug: Sevoflurane + Fentanyl
- IR (Experimental): Sevoflurane (Inhalation)+Remifentanyl
  Interventions: Drug: Sevoflurane + Remifentanyl
- ER (Experimental): Propofol (Endovenous)+ Remifentanyl
  Interventions: Drug: Propofol + Remifentanyl

INTERVENTIONS:
Drug: Sevoflurane + Fentanyl — Sevoflurane is maintained in a MAC range (0.75% to 1.25%) and fentanyl (2-3 microg/kg/hr or 0.7 microg/kg boluses). Just before incision of the scalp, fentanyl (1-2microg/kg/hr) can be supplemented, if necessary
  Arms: IF
Drug: Sevoflurane + Remifentanyl — Sevoflurane is maintained in a MAC range (0.75% to 1.25%) and remifentanil (0.5-0.25 microg/kg/min reduced to 0.05-0.1 microg/kg/min after dural opening). Just before incision of the scalp, remifentanil can be supplemented, if necessary
  Arms: IR
Drug: Propofol + Remifentanyl — Propofol is maintained with continuous infusion at 10 mg/kg/h for the first 10 minutes, then reduced to 8 mg/kg/h for the following 10 minutes and reduced to 6mg/kg/h thereafter and remifentanil 0.5-0.25 microg/kg/min reduced to 0.05-0.1 microg/kg/min after dural opening. Just before incision of the scalp, remifentanil could be supplemented, if necessary
  Arms: ER

SUMMARY:
This protocol, NeuroMorfeo, aims to assess equivalence between volatile and intravenous anesthetics for neurosurgical procedures.

DETAILED DESCRIPTION:
NeuroMorfeo is a multicenter, randomized, open label, controlled trial, based on an equivalence design. Patients aged between 18 and 75 years, scheduled for a elective craniotomy for supratentorial lesion without signs of intracranial hypertension, in good physical state evaluated with the ASA (I-III) and Glasgow Coma Scale (GCS) equal to 15, will be randomly assigned to one of three anesthesiological strategies (two VA arms, sevoflurane + fentanyl or sevoflurane + remifentanil, and one IA, propofol + remifentanil). The equivalence between intravenous and volatile-based neuroanesthesia will be evaluated by comparing the intervals required to reach, after anesthesia discontinuation, a modified Aldrete score ≥ 9 (primary end-point). Two statistical comparisons have been planned: 1) sevoflurane + fentanyl vs. propofol + remifentanil; 2) sevoflurane + remifentanil vs. propofol + remifentanil.

Secondary end-points include: an assessment of neurovegetative stress based on (a) measurement urinary catecholamines and plasma and urinary cortisol and (b) estimate of sympathetic/parasympathetic balance by power spectrum analyses of electrocardiographic tracings recorded during anesthesia; intraoperative adverse events (i.e. hypotension, hypertension, requirement of osmotic agents or/and hyperventilation for controlling brain swelling); evaluation of surgical field; postoperative adverse events (as seizures, cough, shivering, agitation, postoperative hematoma and postoperative pain); patient's satisfaction and an analysis of costs.

411 patients will be recruited in 14 different Italian centers during an 18-month period.

The recruitment started December 20th, 2007 and up to 11th March 2009.

ELIGIBILITY:
Inclusion criteria:

* Patient scheduled for elective intracranial surgery under general anesthesia for a supratentorial mass lesion in the next 24 hours;
* Physical state, evaluated with the ASA (American Society of Anesthesiologists ) classification I (normal healthy patient), II (patient with mild systemic disease), or III (patient with severe systemic disease);
* Age 18-75 years;
* Normal preoperative level of consciousness, i.e. Glasgow Coma Scale (GCS) = 15;
* No signs of intracranial hypertension.

Exclusion criteria:

* Severe cardiovascular pathology, as uncontrolled arterial hypertension, documented reduced coronary reserve.
* Renal or liver disease precluding the use of either anesthetic technique.
* Pregnancy .
* Known allergies to any anesthetic agent.
* Reduced preoperative level of consciousness, i.e.
* Glasgow Coma Scale (GCS) < 15.
* Body weight greater than 120 kg.
* History of drug abuse or psychiatric conditions.
* Documented disturbance of the hypothalamic region.Refusal to sign consent form.
* Participation in other clinical trials.
* Delayed awakening, because, due to the location or size of the lesion, postoperative sedation and mechanical ventilation are planned.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Post-anesthesia awaking time, assessed as the interval (min:sec)required to reach an ALDRETE score ≥ 9 | From estubation to aldrete score ≥ 9

SECONDARY OUTCOMES:
Neurovegetative stress | From induction of anesthesia to 24 hours after surgery
Intraoperative and post-operative adverse events assessment | From induction of anesthesia to 24 hours after surgery
Brain relaxation evaluated by a blinded neurosurgeon | From induction of anesthesia to 24 hours after surgery
Patient's satisfaction | From induction of anesthesia to 24 hours after surgery
Costs of the three strategies | From induction of anesthesia to end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, MD, Principal Investigator — Azienda Ospedaliera San Gerardo Monza; Antonio Pesenti, MD, Study Chair — Università delgi Studi Milano Bicocca; Maria Grazia Franzosi, PhD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri; Roberto Latini, MD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (15):
- Italy (15):
  - Policlinico Consorziale di Bari, Bari
  - Ospedale Bellaria Bologna, Bologna
  - IRCCS Fondazione San Raffaele Milano, Milan
  - Istituto di Ricerche Farmacologiche Mario Negri - Dipartimento di Ricerca Cardiovascolare-, Milan
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale Maggiore della Carità di Novara, Novara
  - Ospedale di Padova, Padua
  - Azienda Ospedaliera di Parma, Parma
  - Policlinico "A. Gemelli" Roma, Rome
  - Policlinico "Umberto I" Roma, Rome
  - Azienda Universitaria Senese, Siena
  - Ospedale San Giovanni Bosco Torino, Turin
  - Ospedale San giovanni Battista Torino, Turin
  - Ospedale di Circolo e Fondazione Macchi Varese, Varese
  - Azienda Ospedaliera Universitaria di Verona, Verona

REFERENCES:
- [Background] Hans P, Bonhomme V. Why we still use intravenous drugs as the basic regimen for neurosurgical anaesthesia. Curr Opin Anaesthesiol. 2006 Oct;19(5):498-503. doi: 10.1097/01.aco.0000245274.69292.ad. PMID 16960481
- [Background] Todd MM, Warner DS, Sokoll MD, Maktabi MA, Hindman BJ, Scamman FL, Kirschner J. A prospective, comparative trial of three anesthetics for elective supratentorial craniotomy. Propofol/fentanyl, isoflurane/nitrous oxide, and fentanyl/nitrous oxide. Anesthesiology. 1993 Jun;78(6):1005-20. doi: 10.1097/00000542-199306000-00002. PMID 8512094
- [Background] Engelhard K, Werner C. Inhalational or intravenous anesthetics for craniotomies? Pro inhalational. Curr Opin Anaesthesiol. 2006 Oct;19(5):504-8. doi: 10.1097/01.aco.0000245275.76916.87. PMID 16960482
- [Background] Magni G, Baisi F, La Rosa I, Imperiale C, Fabbrini V, Pennacchiotti ML, Rosa G. No difference in emergence time and early cognitive function between sevoflurane-fentanyl and propofol-remifentanil in patients undergoing craniotomy for supratentorial intracranial surgery. J Neurosurg Anesthesiol. 2005 Jul;17(3):134-8. doi: 10.1097/01.ana.0000167447.33969.16. PMID 16037733
- [Background] Talke P, Caldwell JE, Brown R, Dodson B, Howley J, Richardson CA. A comparison of three anesthetic techniques in patients undergoing craniotomy for supratentorial intracranial surgery. Anesth Analg. 2002 Aug;95(2):430-5, table of contents. doi: 10.1097/00000539-200208000-00036. PMID 12145066
- [Background] Gomberg-Maitland M, Frison L, Halperin JL. Active-control clinical trials to establish equivalence or noninferiority: methodological and statistical concepts linked to quality. Am Heart J. 2003 Sep;146(3):398-403. doi: 10.1016/S0002-8703(03)00324-7. PMID 12947355
- [Background] Aldrete JA. The post-anesthesia recovery score revisited. J Clin Anesth. 1995 Feb;7(1):89-91. doi: 10.1016/0952-8180(94)00001-k. No abstract available. PMID 7772368
- [Background] Balakrishnan G, Raudzens P, Samra SK, Song K, Boening JA, Bosek V, Jamerson BD, Warner DS. A comparison of remifentanil and fentanyl in patients undergoing surgery for intracranial mass lesions. Anesth Analg. 2000 Jul;91(1):163-9. doi: 10.1097/00000539-200007000-00030. PMID 10866905
- [Background] Del Gaudio A, Ciritella P, Perrotta F, Puopolo M, Lauta E, Mastronardi P, De Vivo P. Remifentanil vs fentanyl with a target controlled propofol infusion in patients undergoing craniotomy for supratentorial lesions. Minerva Anestesiol. 2006 May;72(5):309-19. English, Italian. PMID 16675939
- [Background] Klingstedt C, Giesecke K, Hamberger B, Jarnberg PO. High- and low-dose fentanyl anaesthesia: circulatory and plasma catecholamine responses during cholecystectomy. Br J Anaesth. 1987 Feb;59(2):184-8. doi: 10.1093/bja/59.2.184. PMID 3828169
- [Background] Nishiyama T, Yamashita K, Yokoyama T. Stress hormone changes in general anesthesia of long duration: isoflurane-nitrous oxide vs sevoflurane-nitrous oxide anesthesia. J Clin Anesth. 2005 Dec;17(8):586-91. doi: 10.1016/j.jclinane.2005.03.009. PMID 16427527
- [Background] Desborough JP. The stress response to trauma and surgery. Br J Anaesth. 2000 Jul;85(1):109-17. doi: 10.1093/bja/85.1.109. No abstract available. PMID 10927999
- [Background] Bent JM, Paterson JL, Mashiter K, Hall GM. Effects of high-dose fentanyl anaesthesia on the established metabolic and endocrine response to surgery. Anaesthesia. 1984 Jan;39(1):19-23. doi: 10.1111/j.1365-2044.1984.tb09447.x. PMID 6696213
- [Background] Heesen M, Deinsberger W, Dietrich GV, Detsch O, Boldt J, Hempelmann G. Increase of interleukin-6 plasma levels after elective craniotomy: influence of interleukin-10 and catecholamines. Acta Neurochir (Wien). 1996;138(1):77-80. doi: 10.1007/BF01411728. PMID 8686529
- [Background] Ledowski T, Bein B, Hanss R, Paris A, Fudickar W, Scholz J, Tonner PH. Neuroendocrine stress response and heart rate variability: a comparison of total intravenous versus balanced anesthesia. Anesth Analg. 2005 Dec;101(6):1700-1705. doi: 10.1213/01.ane.0000184041.32175.14. PMID 16301244
- [Background] Guzzetti S, Borroni E, Garbelli PE, Ceriani E, Della Bella P, Montano N, Cogliati C, Somers VK, Malliani A, Porta A. Symbolic dynamics of heart rate variability: a probe to investigate cardiac autonomic modulation. Circulation. 2005 Jul 26;112(4):465-70. doi: 10.1161/CIRCULATIONAHA.104.518449. Epub 2005 Jul 18. PMID 16027252
- [Background] Olsen KS, Pedersen CB, Madsen JB, Ravn LI, Schifter S. Vasoactive modulators during and after craniotomy: relation to postoperative hypertension. J Neurosurg Anesthesiol. 2002 Jul;14(3):171-9. doi: 10.1097/00008506-200207000-00001. PMID 12172288
- [Background] Leslie K, Troedel S. Does anaesthesia care affect the outcome following craniotomy? J Clin Neurosci. 2002 May;9(3):231-6. doi: 10.1054/jocn.2001.0934. No abstract available. PMID 12093125
- [Background] Hall GM, Young C, Holdcroft A, Alaghband-Zadeh J. Substrate mobilisation during surgery. A comparison between halothane and fentanyl anaesthesia. Anaesthesia. 1978 Nov-Dec;33(10):924-30. PMID 727414
- [Background] Fung D, Cohen M, Stewart S, Davies A. Can the Iowa Satisfaction with Anesthesia Scale be used to measure patient satisfaction with cataract care under topical local anesthesia and monitored sedation at a community hospital? Anesth Analg. 2005 Jun;100(6):1637-1643. doi: 10.1213/01.ANE.0000154203.00434.23. PMID 15920188
- [Background] Citerio G, Stocchetti N, Cormio M, Beretta L. Neuro-Link, a computer-assisted database for head injury in intensive care. Acta Neurochir (Wien). 2000;142(7):769-76. doi: 10.1007/s007010070091. PMID 10955671
- [Background] Piper I, Citerio G, Chambers I, Contant C, Enblad P, Fiddes H, Howells T, Kiening K, Nilsson P, Yau YH; BrainIT Group. The BrainIT group: concept and core dataset definition. Acta Neurochir (Wien). 2003 Aug;145(8):615-28; discussion 628-9. doi: 10.1007/s00701-003-0066-6. PMID 14520540
- [Background] Piaggio G, Elbourne DR, Altman DG, Pocock SJ, Evans SJ; CONSORT Group. Reporting of noninferiority and equivalence randomized trials: an extension of the CONSORT statement. JAMA. 2006 Mar 8;295(10):1152-60. doi: 10.1001/jama.295.10.1152. PMID 16522836
- [Background] Le Henanff A, Giraudeau B, Baron G, Ravaud P. Quality of reporting of noninferiority and equivalence randomized trials. JAMA. 2006 Mar 8;295(10):1147-51. doi: 10.1001/jama.295.10.1147. PMID 16522835
- [Background] Kaul S, Diamond GA. Good enough: a primer on the analysis and interpretation of noninferiority trials. Ann Intern Med. 2006 Jul 4;145(1):62-9. doi: 10.7326/0003-4819-145-1-200607040-00011. PMID 16818930
- [Derived] Citerio G, Franzosi MG, Latini R, Masson S, Barlera S, Guzzetti S, Pesenti A. Anaesthesiological strategies in elective craniotomy: randomized, equivalence, open trial--the NeuroMorfeo trial. Trials. 2009 Apr 6;10:19. doi: 10.1186/1745-6215-10-19. PMID 19348675